CLINICAL TRIAL: NCT05701514
Title: The COllaborative Neonatal Network for the First Congenital Pulmonary Airway Malformation (CPAM) Trial
Brief Title: The COllaborative Neonatal Network for the First CPAM Trial
Acronym: CONNECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, dr. J Marco Schnater, dr. J.M. Schnater, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT-study
Record Dates: First submitted 2022-12-15; First posted 2023-01-27 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Congenital Pulmonary Airway Malformation
Keywords: Asymptomatic CPAM; Optimal management; Conservative vs surgical; Randomized
MeSH Terms: conditions — Cystic Adenomatoid Malformation of Lung, Congenital | interventions — Aging

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, multicentre superiority trial. Randomisation will take place as blocked randomisation with stratification by centre, with a 1:1 allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative arm (No Intervention): Children assigned to this treatment arm will be conservatively managed, and will continue to be followed until the age of 5 years (end of study inclusion).
- Surgical arm (Active Comparator): Children assigned to this treatment arm will undergo elective surgical resection at the age of 6-9 months, and will continue to be followed until the age of 5 years (end of study inclusion).
  Interventions: Procedure: Elective surgical resection of CPAM between 6 and 9 months of age

INTERVENTIONS:
Procedure: Elective surgical resection of CPAM between 6 and 9 months of age — Surgical resection of the CPAM between 6 and 9 months of age
  Arms: Surgical arm

SUMMARY:
The goal of this clinical trial is to compare conservative wait-and-see management to elective surgical intervention, in asymptomatic Congenital Pulmonary Airway Malformation (CPAM) children.

Children assigned to the intervention group will undergo surgical resection of the CPAM between 6 and 9 months of age. Children assigned to the control group will be monitored conservatively. The follow-up scheme will be uniform for both treatment groups and last for 5 years.

The primary outcome is the difference in maximal endurance at five years of age between the surgical and conservative group. Secondary outcome measures are molecular genetic diagnostics, validated questionnaires - on parental anxiety, quality of life and health care consumption -, repeated imaging, and pulmonary morbidity during follow-up, as well as surgical complications and histopathology.

DETAILED DESCRIPTION:
Study design: prospective multicentre randomized controlled trial. Duration: the total duration of the follow-up will be 5 years Setting: collaborating centres within the COllaborative Neonatal Network for the first European Congenital Pulmonary Airway Malformation (CPAM) Trial consortium (CONNECT)

Parents expecting a child with a prenatally diagnosed CPAM will be counselled and informed about the study prenatally. At the age of 6 months, each child will undergo a chest CT with intravenous contrast in order to confirm the diagnosis, as part of the standard of care. This chest CT will be evaluated according to a structured report. If the chest CT confirms the diagnosis CPAM and the child remains asymptomatic, the child is eligible for inclusion. After having obtained informed consent from parents or caregivers, randomisation to the surgical arm or the non-surgical arm will take place. At this point, the prenatal ultrasound images will be retrospectively evaluated according to a structured report.

In case of randomisation to the surgical arm, surgical resection will take place between 6 and 9 months of age. The type and extent of the surgical procedure is dependent on the lesion characteristics, local protocol and the surgeon's preference. Preferably, small lesions are treated with a segmentectomy; i.e., sub-lobar resection. Larger lesions are generally treated with lobectomy. Wedge resection is not advised due to higher risks of post-operative air leakage and residual disease. Surgical details will be documented according to a structured report.

Resected material will be sent to the local pathology department for analysis. The local pathologist will analyse the material, and document the results according to the Structured Pathology Report for Congenital Pulmonary Airway Malformation.

Genetic testing will be offered as part of routine diagnostic procedures. Standard information leaflets and informed consent forms of the department of clinical genetics will be offered to parents. If parental consent is obtained, blood (1-4ml, depending on availability/safety) will be drawn from the study subject, at the moment when an IV-needle is placed - in order to administer the IV-contrast - just before the diagnostic CT-scan). This material will be stored in a plastic Etheylenediaminetetraacetic acid (EDTA) vacutainer blood collector tube. Similarly, blood of both parents - if possible - (10 ml) will be drawn and stored in a plastic EDTA vacutainer blood collector tube. These parental samples will be sent for DNA isolation and genetic analysis to the local departments of Clinical Genetics, where the DNA will be stored. In this diagnostic procedure, trio single nucleotide polymorphism (SNP) array / whole exome sequencing or whole genome sequencing will be performed.

The follow-up program lasts 5 years, is uniform for all patients and consists of three assessments at the ages of 1 year, 2.5 years, and 5 years (with a margin of 2 months towards the patients' age for each assessment). This follow-up structure is standard of care in the majority of the participating centres. Patients assigned to the surgical arm will visit the hospital one additional time, 2-6 weeks after the surgery has taken place, for scar inspection, postoperative complaints and evaluation of the pathology report. At the second visit (at 2.5 years) a follow-up CT-scan will be performed, and during the last visit participants will perform a standardised exercise test using the BRUCE treadmill protocol, supervised by a certified paediatric physical therapist.

Furthermore, parents will be asked to complete several questionnaires, addressing anxiety, quality of life and medical costs.

The duration of the follow-up was set to 5 years to ensure enough time to observe potential differences in clinical outcome between the two study groups (i.e., the development of post-surgical complications or the development of symptoms in the conservative group). Another consideration was that the age of 5 years is the youngest age at which standardised endurance tests have been validated.

ELIGIBILITY:
Inclusion Criteria:

* Lesion detected during routine prenatal ultrasound screening
* Delivery at term: gestational age ≥37 weeks
* Birthweight > -2SD or >P10
* Asymptomatic at birth defined as no prolonged respiratory distress or oxygen support (< 24 hours)
* Asymptomatic up to the moment of inclusion
* Confirmation of CPAM on postnatal chest CT-scan at 3-9 months of age, according to structured report form (34)
* Unilateral lesion occupying no more than one lung lobe as assessed on chest CT-scan at 3-9 months of age

Exclusion Criteria:

* Bilateral lesion
* Development of symptoms before randomization, considered by treating physician as caused by CPAM with reasonable certainty
* Complicated pregnancy defined as (pre-)eclampsia, pregnancy diabetes in mother, foetal hydrops or severe polyhydramnios on prenatal ultrasound
* Syndrome associated anomalies on genetic analysis confirmed by genetic expert
* Major associated malformations. Anomalies include cardiac malformations requiring surgical correction or follow-up by a paediatric cardiologist, congenital malformations requiring major surgical intervention, and anomalies that affect normal lung growth and development.
* Suspicion of malignancy on chest CT scan evaluation at the age of 3-9 months
* Participation in another randomised controlled trial

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Exercise tolerance | 5 years
  BRUCE treadmill test protocol. Total endurance time will be converted to a sex and age matched percentile score based on pre-defined reference values.

SECONDARY OUTCOMES:
Pulmonary morbidity during follow-up | through study completion, a total of 5 years
  Infection, cough, dyspea, respiratory insufficiency etc.
Surgical intervention due to pulmonary morbidity | Through study completion, a total of 5 years
  Indication for surgical resection of the pulmonary lesion following the development of pulmonary morbidity during follow-up
CPAM characteristics on prenatal ultrasound images, according to standardized structured report | 20 weeks gestation
  Structured report form to be added up to 1 score, in which case a higher score indicates a larger and more complicated lesion
CPAM characteristics on postnatal CT-scan, according to standardized structured report | 3-9 months of age
  Structured report form to be added up to 1 score, in which case a higher score indicates a larger and more complicated lesion
CPAM development / post-surgical appearance on repeated CT imaging, according to standardized structured report | 2.5 years of age
  Structured report form to be added up to 1 score, in which case a higher score indicates a larger and more complicated lesion
CPAM development / post-surgical appearance on CT imaging - scored according to the Congenital Lung Abnormalities Quantification (CLAQ) method | 3-9 months of age + 2.5 years of age
  Structured report form to be added up to 1 score, in which case a higher score indicates a larger and more complicated lesion
Quality of life analysis | 6 months, 1 year, 2.5 years, 5 years
  Toddler Quality of Life Questionnaire (ITQOL), transformed to a scale score from 0 (worst health) to 100 (best health)
Quality of life analysis | 5 years
  Child Health Utility Index (CHU9D). Translated to total raw scores ranging from 0 (no impairment) to 36 (maximal impairment) based 9 questions in 9 different dimensions.
Parental anxiety level, assessed pre-operatively | 6 months, 1 year, 2.5 years, 5 years
  Visual Analogue Scale for Anxiety (VAS-A), scored from 0 (no anxiety) to 10 (maximal anxiety).
Weight | 6 months, 1 year, 2.5 years, 5 years
  Converted to Standard Deviation score
Height | 6 months, 1 year, 2.5 years, 5 years
  Converted to Standard Deviation score
Pathological characteristics of resected material, according to standardized structured report | 9-12 months
  Structured report form to be added up to 1 score, in which case this score defines specific, pre-defined pathological lesion characteristics. This score does therefore not indicate better of worse, but rather specifies the lesion characteristics.
Cost-effectiveness of both management strategies and comparison | 6 months, 1 year, 2.5 years, 5 years
  The cost consequences and cost-effectiveness of surgical versus conservative management of CPAM will be analyzed through a trial-based economic evaluation.
  Data on health care resource consumption will be extracted from both the electronic information systems of the participating centres and the Institute for Medical Technology Assessment (iMTA) Medical Consumption Questionnaire (iMCQ).
  As regards the effects of the intervention, the economic evaluation will look at maximal endurance time and quality-adjusted life-years (QALYs), which is a measure of health outcome that combines quality of life with length of life. The calculation of QALYs will be based on survival data and on responses to the Child Health Utility 9D (CHU9D) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rene MH Wijnen, professor, Study Director — Head of department Pediatric Surgery, Erasmus MC Sophia Children's Hospital, Rotterdam
Locations (2):
- Netherlands (2):
  - Radboud University Medical Centre, Nijmegen, Gelderlanf
  - Erasmus MC Sophia Children's Hospital, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: Open access

REFERENCES:
- [Background] Hermelijn S, Kersten C, Mullassery D, Muthialu N, Cobanoglu N, Gartner S, Bagolan P, Mesas Burgos C, Sgro A, Heyman S, Till H, Suominen J, Schurink M, Desender L, Losty P, Ertresvag K, Tiddens HAWM, Wijnen RMH, Schnater M; CONNECT study consortium COS development group; CONNECT study consortium COS development group. Development of a core outcome set for congenital pulmonary airway malformations: study protocol of an international Delphi survey. BMJ Open. 2021 Apr 12;11(4):e044544. doi: 10.1136/bmjopen-2020-044544. PMID 33846152
- [Background] Kersten CM, Hermelijn SM, Mullassery D, Muthialu N, Cobanoglu N, Gartner S, Bagolan P, Mesas Burgos C, Sgro A, Heyman S, Till H, Suominen J, Schurink M, Desender L, Losty P, Steyaert H, Terheggen-Lagro S, Metzelder M, Bonnard A, Sfeir R, Singh M, Yardley I, Rikkers-Mutsaerts NRVM, van der Ent CK, Qvist N, Cox DW, Peters R, Bannier MAGE, Wessel L, Proesmans M, Stanton M, Hannon E, Zampoli M, Morini F, Tiddens HAWM, Wijnen RMH, Schnater JM. The Management of Asymptomatic Congenital Pulmonary Airway Malformation: Results of a European Delphi Survey. Children (Basel). 2022 Jul 30;9(8):1153. doi: 10.3390/children9081153. PMID 36010044
- [Derived] Kersten CM, Hermelijn SM, Dossche LWJ, Muthialu N, Losty PD, Schurink M, Rietman AB, Poley MJ, van Rosmalen J, Zanen-van den Adel TPL, Ciet P, von der Thusen J, Brosens E, Ijsselstijn H, Tiddens HAWM, Wijnen RMH, Schnater JM. COllaborative Neonatal Network for the first European CPAM Trial (CONNECT): a study protocol for a randomised controlled trial. BMJ Open. 2023 Mar 17;13(3):e071989. doi: 10.1136/bmjopen-2023-071989. PMID 36931672